CLINICAL TRIAL: NCT02485717
Title: A Phase 3, Randomized, Double Blind, Placebo-Controlled Study to Assess the Safety, Efficacy and Pharmacokinetics of Natroba™ (Spinosad) for the Treatment of Scabies
Brief Title: Phase 3 Trial to Assess the Safety and Efficacy of Natroba for the Treatment of Scabies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ParaPRO LLC (Industry)
Collaborators: Concentrics Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPN-303-15
Record Dates: First submitted 2015-06-19; First posted 2015-06-30 (Estimated); Results first posted 2019-01-16 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-04

CONDITIONS: Scabies
MeSH Terms: conditions — Scabies | interventions — spinosad; Suspensions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Natroba (spinosad) (Experimental): spinosad topical suspension, 0.9% up to 120 mL (enough product is used to cover the body from the neck down to the soles of the feet), one treatment left on for 6 hours
  Interventions: Drug: spinosad topical suspension, 0.9%
- Placebo (Placebo Comparator): placebo is a topical suspension that is the same formulation as Natroba without the active ingredient spinosad. Up to 120 mL (enough product is used to cover the body from the neck down to the soles of the feet), one treatment left on for 6 hours.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: spinosad topical suspension, 0.9% — Topically apply 0.9% suspension up to 120 mL (enough to cover the body from the neck down to the soles of the feet). One application for six hours.
  Other Names: Natroba (spinosad) Topical Suspension, 0.9%
  Arms: Natroba (spinosad)
Other: Placebo — Placebo is the same as the drug minus the active ingredient spinosad (vehicle). Topically apply up to 120 mL (enough to cover the body from the neck down to the soles of the feet). One application for six hours.
  Arms: Placebo

SUMMARY:
To assess the safety and efficacy of Natroba (spinosad) topical suspension versus placebo for the clinical cure of scabies after a single treatment. The trial will also assess the pharmacokinetics (PK) of spinosad and benzyl alcohol following a single dose of Natroba™ in pediatric subjects 4-16 years of age. These subjects will be a separate population of pediatric subjects.

DETAILED DESCRIPTION:
The primary study is a double blind, two-arm, 28-day, placebo-controlled study with approximately 120 infested "index" subjects randomized 1:1 to Natroba™ or Placebo. All members of a household (no more than 6 individuals) with a suspected "index" subject must be screened at the first visit. In this study, "index" subjects are defined as the youngest infested household member (≥4 years). If the members have an active scabies infestation and meet all other criteria, they must agree to participate in the study. Household members who do not present with scabies at the screening visit must also agree to apply the same blinded investigational product (IP) as household members who present with scabies. All household members must agree to participate in the study or none will be enrolled. Screening procedures include informed consent, medication and medical history, urine pregnancy test for females of childbearing potential, scabies assessment (visual evidence of burrows, inflammatory/non-inflammatory lesions and pruritus), microscopic examination of skin scraping, or dermatoscopy, to demonstrate the presence of mites, eggs, and/or scybala (dermatoscopy must confirm burrows), vital signs, general skin and eye assessment, randomization, CBC and serum chemistry, and IP dispensing and instruction.

After screening on Day 1, all randomized subjects in the primary population will be dispensed IP (Natroba™ or Placebo) to apply at home later the same day as a single treatment over the entire body from the neck down to the toes (including the soles of the feet) and to the scalp (if balding) or hairline, temples and forehead on the same day. Subjects less than 12 years of age should be assisted with administration by a parent, guardian or caregiver. Subjects will rub the treatment into the skin followed by a 10-minute wait period before getting dressed. Showering or bathing must not occur earlier than 6 hours after treatment and no later than at least 1 hour prior to Day 2 visit.

A separate population of 24 pediatric "non-index" subjects that do not reside in the "index" subject's household will be enrolled to assess the PK of spinosad and benzyl alcohol for 12 hours after open-label topical application on a single in-clinic visit (Day 1, or Day 2 if screening only on Day 1). There will be 12 male or female subjects 4 - 9 years of age (with a minimum of 6 male or female subjects 4 - 6 years of age) and 12 male or female subjects 10 - 16 years of age. With assistance from a caregiver, Natroba™ will be applied over entire body from the neck down to the toes (including the soles of the feet) and to the hairline, temples, and forehead. The open-label product will remain on the skin for at least 6 hours before bathing or showering. The subjects will stay in the clinic until the 12-hour procedures are completed. Blood draws will be taken at 0 hours just prior to treatment, and then at 0.5, 1.0, 3.0, 6.0 hours post-treatment and then at 12 hours post-treatment. Bathing must occur after the 6 hour blood draw but prior to the 12 hour blood draw. A ±5 minute time window will be allowed for all post-treatment blood samples. Safety will be assessed with adverse events (AEs), general skin and eye irritation assessments, pre-dose and pre-discharge laboratory evaluations, and vital signs during the 12 hours in-clinic. Following the sample collections subjects will be released from the clinic and directed to their primary care physician for follow-up. PK subjects will be provided 5% Permethrin upon discharge to dispense to household members.

In the primary population (all household members), on Day 2 (Visit 2), general skin and eye assessments will be made for possible irritation, and to confirm that all IP was left on for a minimum of 6 hours before bathing or showering. If a subject reports an adverse event assessed as related by the PI on Day 2 (Visit 2) then a follow-up visit with the investigator must be scheduled within 7 days of visit. Subjects will receive a well-being phone call on Day 14 to continue to emphasize instructions to prevent re-infestation, determine if any concomitant medications have been used, and check for adverse events. If a subject reports an adverse event assessed as related by the PI on the Day 14 well-being phone call, then a follow-up visit with the investigator must be scheduled within 7 days of phone call.

On Day 28 (Visit 3), all household members will return to the clinic for safety and efficacy assessments. The primary endpoint of complete cure will be assessed in the infested household members. If the infested subject is completely cured at Day 28, he or she will have completed the study and termination procedures will be conducted. If the subject is not completely cured at Day 28 (with Natroba™ or Placebo), the subject will receive 5% Permethrin and will be directed to their primary care physician for follow-up.

Safety assessments will be made for all household members and will include monitoring of adverse events (AEs) throughout the study, vital signs recording (Days 1 and 28), clinical laboratory analyses (Days 1 and 28), and general skin and eye irritation assessments (Days 1, 2, and 28).

The Day 28 procedures will also be completed for early termination (ET) except subjects will not receive rescue Permethrin, but will be directed to follow-up with their primary care physician.

ELIGIBILITY:
Inclusion Criteria:

* All household members who have provided written informed consent and an authorization for disclosure of protected health information must meet all the following criteria:

  1. Male or female, age 4 years and upward.
  2. At least one household member must have active scabies infestation confirmed by clinical signs and symptoms (evidence of burrows or presence of scabies inflammatory/non-inflammatory lesions and pruritus) as well as by microscopic examination of skin scraping, or dermatoscopy, to demonstrate the presence of mites, eggs, and/or scybala. If dermatoscopy is used it should also confirm there are burrows on the skin.
  3. Generally in good health based on medical history and clinical assessments.
  4. Normal-appearing skin in noninfested areas.
  5. No history of chronic or recurrent dermatologic disease.
  6. Willingness to comply with the study procedures including blood collections and application of study treatment at home or in-clinic (PK subjects).
  7. Willing and able to practice an acceptable measure of contraception during the study, if female of childbearing potential. Examples of acceptable contraceptive methods include abstinence, intrauterine device (IUD) or double barrier method, oral or injectable contraceptives (must have been using consistent systemic contraceptives for at least 3 months prior to enrollment). If abstinent and planning to become sexually active with a household member must agree to use a double barrier method.
  8. Subject agrees to inform their sexual partners to seek an examination for scabies and treatment if, and when, symptoms present.
  9. Household members must be 6 or fewer and all members must be willing to attend clinic visits and be randomized to treatment (blinded, but same for all).

Exclusion Criteria:

* All household members must be excluded if any of the following conditions are met:

  1. Household has greater than 6 residents.
  2. Has a household member(s) who is not willing or not eligible to enroll.
  3. Presence of scabies on the scalp.
  4. Presence of crusted scabies (Norwegian scabies).
  5. Allergies or intolerance to ingredients in the IPs.
  6. Current pregnancy (as assessed by urine pregnancy test) or currently nursing.
  7. The household has sexually active subjects who do not agree to restrict prolonged skin to skin contact with non-household members during the trial period.
  8. Known renal or hepatic impairment.
  9. Treatment with scabicide within the prior 4 weeks.
  10. Immunodeficiency (including HIV infection) as reported in Medical History.
  11. Signs or symptoms of systemic infection.
  12. Administration of systemic therapy for infectious disease within the prior 2 weeks.
  13. Receipt of any IP within the prior 4 weeks.
  14. Any other conditions that, at the investigator's discretion, may interfere with the study conduct, or which might confound the interpretation of the study results, or which may put the subject at undue risk.
  15. Does not have a known household affiliation with their household members (stays in one household inconsistently, i.e., sleeps at one place several nights and then other places on other nights).
  16. Household member is unwilling to treat scabies.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 291 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2018-06-25 (Actual); Study Completion 2018-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kerry W Mettert, MBA, Study Director — ParaPRO LLC
Locations (5):
- United States (5):
  - Elk Grove Clinical Research, Elk Grove, California
  - The Chappel Group Research, Kissimmee, Florida
  - San Marcus Research, Miami, Florida
  - L&C Professional Medical Research Institute, Miami, Florida
  - LSRN Research, West Palm Beach, Florida

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Exclusion Criteria #2 - Has a household member(s) who is not willing or not eligible to enroll.
  Exclusion Criteria #12 - Administration of systemic therapy for infectious disease within the prior 2 weeks.
Groups:
- PK Natroba (Spinosad): open-label spinosad topical suspension, 0.9% up to 120 mL (enough product is used to cover the body from the neck down to the soles of the feet), one treatment left on for 6 hours
  open-label spinosad topical suspension, 0.9%: Topically apply 0.9% suspension up to 120 mL (enough to cover the body from the neck down to the soles of the feet). One application for six hours.
Period: Overall Study
Arm/Group | Natroba (Spinosad) | Placebo | PK Natroba (Spinosad)
Started | 142 | 129 | 20
Completed | 136 | 127 | 19
Not Completed | 6 | 2 | 1
Not completed — Lost to Follow-up | 6 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Did Not Meet Exclusion Criteria #2 | 0 | 1 | 0
Not completed — Did Not Meet Exclusion Criteria #12 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Natroba (Spinosad) | Placebo | PK Natroba (Spinosad) | Total
Number analyzed (Participants) | 142 | 129 | 20 | 291
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30 | 35 | 20 | 85
  Between 18 and 65 years | 94 | 82 | 0 | 176
  >=65 years | 18 | 12 | 0 | 30
Age, Continuous [Mean (Full Range); unit: Years] | 38.7 [5 to 89] | 38.4 [4 to 83] | 9.6 [5 to 16] | 36.5 [4 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 70 | 8 | 151
  Male | 69 | 59 | 12 | 140
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 2
  Black or African American | 11 | 7 | 4 | 22
  White | 130 | 121 | 15 | 266
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 142 | 129 | 20 | 336
Evidence of Burrows [Count of Participants; unit: Participants] | 38 | 42 | 6 | 86
Evidence of Lesions [Count of Participants; unit: Participants] | 63 | 69 | 20 | 152
Evidence of Pruritus [Count of Participants; unit: Participants] | 71 | 75 | 20 | 166
Total Number of Pre-existing Lesions [Mean (Full Range); unit: lesions] | 10.8 [0 to 150] | 11.3 [0 to 100] | 12.0 [3 to 34] | 11.1 [0 to 150]
Score of Pre-existing Lesions [Count of Participants; unit: Participants]
  Free of Lesions | 79 | 60 | 0 | 139
  ≤ 10 Lesions (Mild) | 20 | 26 | 11 | 57
  11-49 Lesions (Moderate) | 40 | 37 | 9 | 86
  ≥ 50 Lesions (Severe) | 3 | 6 | 0 | 9
Microscopic/Dermatoscopy Result [Count of Participants; unit: Participants]
  Negative | 73 | 59 | 0 | 132
  Positive | 63 | 68 | 20 | 151
  Not Done | 6 | 2 | 0 | 8
Active Scabies Infestation [Count of Participants; unit: Participants] | 63 | 68 | 20 | 151
Prior Scabies Infestation [Count of Participants; unit: Participants] | 28 | 32 | 0 | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Index Subjects Completely Cured of Scabies After a Single Treatment
Description: The primary efficacy assessment is the proportion of index subjects completely cured of scabies by Day 28. Complete cure is defined as a demonstration of both clinical cure (all signs and symptoms have completely resolved, including burrows, inflammatory/non-inflammatory lesions and pruritus) and microscopic or dermatoscopic cure demonstrating the absence of mites, eggs, and/or scybala, and a negative dermatoscopy for burrows.
Time Frame: 28 days after treatment
Population: Participants analyzed are based on the number of subjects who had no missing observations in each study group.
Measure: Count of Participants; unit: Participants
Arm/Group | Natroba (Spinosad) | Placebo
Number analyzed (Participants) | 43 | 43
Participants | 30 | 20

2. Secondary Outcome: This Assessment Includes Assessing the Cmax (μg/mL) of Benzyl Alcohol Pre-dose and During 12 Hours Post-dose of Natroba™ in Pediatric Subjects (Ages 4-16 Years).
Time Frame: 12 Hours
Measure: Mean (Standard Deviation); unit: μg/mL
Groups:
- Pharmacokentic Study: Approximately 24 unique pediatric subjects participated in the PK study. The PK study included approximately 12 male or female subjects aged 4 to 9 years, with a minimum of 6 male or female subjects aged 4 to 6 years; and 12 male or female subjects aged 10 to 16 years. Natroba was applied at the study center during a single visit (Day 1 or Day 2 [only if screening assessments were completed on Day 1]) with assistance from a caregiver according to the same instructions and time restrictions as described for the primary study. Blood samples were collected at 0 hours (just prior to treatment), and then at 0.5, 1.0, 3.0, 6.0, and 12 hours post-treatment (with a ± 5-minute window for each post-treatment time point). The subjects remained at the study center until the 12-hour procedures were completed. Bathing must have occurred after the 6-hour blood draw but prior to the 12-hour blood draw.
Arm/Group | Pharmacokentic Study
Number analyzed (Participants) | 19
μg/mL | 2.737 (1.107)

3. Secondary Outcome: This Assessment Includes Assessing the Tmax (Hours) of Benzyl Alcohol Pre-dose and During 12 Hours Post-dose of Natroba™ in Pediatric Subjects (Ages 4-16 Years).
Time Frame: 12 Hours
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Pharmacokentic Study
Number analyzed (Participants) | 19
hours | 1.42 (1.242)

4. Secondary Outcome: This Assessment Includes Assessing the AUC 0-12h (μg•h/mL) of Benzyl Alcohol Pre-dose and During 12 Hours Post-dose of Natroba™ in Pediatric Subjects (Ages 4-16 Years).
Time Frame: 12 Hours
Measure: Mean (Standard Deviation); unit: μg•h/mL
Arm/Group | Pharmacokentic Study
Number analyzed (Participants) | 19
μg•h/mL | 19.240 (0)

5. Secondary Outcome: This Assessment Includes Assessing the Cmax (ng/mL) of Spinosad (Spinosyn A and Spinosyn D) Pre-dose and During 12 Hours Post-dose of Natroba™ in Pediatric Subjects (Ages 4-16 Years).
Description: Note: All of the spinosad (spinosyn A and spinosyn D) plasma levels tested were below the limit of quantification (3 ng/mL). Therefore, the mean and standard deviation of Cmax read "0" in the Outcome Measure Data Table.
Time Frame: 12 Hours
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Pharmacokentic Study
Number analyzed (Participants) | 19
ng/mL | 0 (0)

6. Secondary Outcome: This Assessment Includes Assessing the Tmax (Hours) of Spinosad (Spinosyn A and Spinosyn D) Pre-dose and During 12 Hours Post-dose of Natroba™ in Pediatric Subjects (Ages 4-16 Years).
Description: Note: All of the spinosad (spinosyn A and spinosyn D) plasma levels tested were below the limit of quantification (3 ng/mL). Therefore, the mean and standard deviation of Tmax read "0" in the Outcome Measure Data Table.
Time Frame: 12 Hours
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Pharmacokentic Study
Number analyzed (Participants) | 19
hours | 0 (0)

7. Secondary Outcome: This Assessment Includes Assessing the AUC 0-12h (ng•h/mL) of Spinosad (Spinosyn A and Spinosyn D) Pre-dose and During 12 Hours Post-dose of Natroba™ in Pediatric Subjects (Ages 4-16 Years).
Description: Note: All of the spinosad (spinosyn A and spinosyn D) plasma levels tested were below the limit of quantification (3 ng/mL). Therefore, the mean and standard deviation of AUC 0-12h read "0" in the Outcome Measure Data Table.
Time Frame: 12 Hours
Measure: Mean (Standard Deviation); unit: ng•h/mL
Arm/Group | Pharmacokentic Study
Number analyzed (Participants) | 19
ng•h/mL | 0 (0)

ADVERSE EVENTS:
Time Frame: 1 year, 1 month
Arm/Group | Natroba (Spinosad) | Placebo | PK Natroba (Spinosad)
All-Cause Mortality (participants affected / at risk) | 0/142 | 0/129 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/142 | 0/129 | 0/20
Other Adverse Events (participants affected / at risk) | 0/142 | 0/129 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site may not publish or publicly present Study results. If Sponsor has given its prior written consent to the Site to publish or present Study results, Site will provide Sponsor with a copy of any proposed oral or written publication to at least sixty (60) days in advance of submission for publication or presentation for review and comment on the appropriateness of the data analysis and presentation. The terms of this paragraph shall survive expiration or termination of this Agreement.

DOCUMENTS (2):
  • Study Protocol (2018-03-23): https://cdn.clinicaltrials.gov/large-docs/17/NCT02485717/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-24): https://cdn.clinicaltrials.gov/large-docs/17/NCT02485717/SAP_001.pdf